CLINICAL TRIAL: NCT00433940
Title: Immune Suppression of Infants Treated With Oral Corticosteroids for Infantile Hemangiomas: A Pilot Study
Brief Title: Immune Suppression Of Infants Treated With Steroids
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Beth Drolet, MD, Medical College of Wisconsin
Other Study IDs: Immune Suppression of Infants
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Hemangioma
Keywords: Hemangioma; Corticosteroid; Prednisone
MeSH Terms: conditions — Hemangioma | interventions — Prednisolone; Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Collection of blood samples at each visit. Following laboratory testing, no samples were retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infantile Hemangioma Patients: Infants with infantile hemangioma being treated clinically with oral prednisolone sodium phosphate suspensions.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Oral prednisolone sodium phosphate suspension administered in dosage of 15mg/5mL. Medication administered every morning at a starting daily dose of 2.5mg/kg.
  Other Names: steroid

SUMMARY:
The goal of this study is to clarify the degree of immune suppression in infants requiring therapy and to create guidelines for evaluation and prevention of infection in infants on oral steroids for hemangiomas.

DETAILED DESCRIPTION:
Infants with large or complicated hemangiomas are often treated systemically with oral steroids. The side effects of the drug on young infants has not been studied. The goal of this study is to clarify the degree of immune suppression in infants requiring therapy and to create guidelines for evaluation and prevention of infection in infants on oral steroids for hemangiomas. Prednisone will be started according to established standard of care. Visits will occur every four weeks for follow-up. There will be six blood draws from baseline to completion of study. Approximately up to 1 ½ teaspoons per blood sample will be drawn to test the strength of the infant's immune system. Participation in this study will last up to 14 months or until stabilization of the hemangioma. Evaluation will occur 12 weeks after discontinuing the steroid for its long-term effects on the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 6 months of age with infantile hemangiomas requiring treatment with oral corticosteroids
* Infant must be enrolled prior to initiation of steroid therapy

Exclusion Criteria:

* Infants > 6 months of age
* Infants already receiving oral corticosteroid treatment prior to the start of this study
* Infants with know immunodeficiencies
* Infants receiving other oral medications for the treatment of hemangiomas

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects were recruited from a hospital based pediatric dermatology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Lymphocyte Subtest of Complete Blood Count Analysis (Primary Immunodeficiency) | 2 years
  Measurement of absolute lymphocyte count and % lymphocyte found during a Complete Blood Count analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Drolet, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States